CLINICAL TRIAL: NCT06079684
Title: Clinical Evidence Regarding The Dynamic of Baker Cyst Dimensions After Intermittent Vacuum Therapy As Rehabilitation Treatment In Patients With Knee Osteoarthritis
Brief Title: Baker Cyst Dimensions and Intermittent Vacuum Therapy in Knee Osteoarthritis (BCIVT)
Acronym: BCIVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balnear and Rehabilitation Sanatorium Techirghiol (Other)
Responsible Party: Principal Investigator, Elena-Valentina Ionescu, Assit. Prof. Dr. Ionescu Elena Valentina, Balnear and Rehabilitation Sanatorium Techirghiol
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BalnearRehabTechirghiol
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Baker Cyst; Knee Osteoarthritis
Keywords: Baker Cyst; Intermittent Vacuum; Knee Osteoarthritis; Ultrasonography; Physical therapy; Mud; Rehabilitation
MeSH Terms: conditions — Popliteal Cyst; Osteoarthritis, Knee | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vacuum Group (Experimental): Vacuum Group with 32 patients: for 10 consecutive days, all patients performed the same program procedures: Intermittent vacuum therapy (for 30 minutes, with a Vacumed device -the lower body was positioned in the vacuum chamber, which was sealed around the participant's trunk with a cuff at the level of the umbilicus to allow application of negative pressure), general warm mud bath (20 minutes at 38 degrees Celsius), hydrokinetotherapy in saline water from Lake Techirghiol by a certified physical therapist (20 minutes at 35 degrees Celsius), massage therapy for paravertebral muscles, shoulder and pelvis girdle and kinesiotherapy with a standard program for peripheric joints for 30 minutes
  Interventions: Device: Intermittent vacuum therapy
- Control Group (Active Comparator): Control Group with 33 patients: for 10 consecutive days, all patients performed the same program procedures: general warm mud bath (20 minutes at 38 degrees Celsius), hydrokinetotherapy in saline water from Lake Techirghiol by a certified physical therapist (20 minutes at 35 degrees Celsius), massage therapy for paravertebral muscles, shoulder and pelvis girdle and kinesiotherapy with a standard program for peripheric joints for 30 minutes
  Interventions: Device: Intermittent vacuum therapy

INTERVENTIONS:
Device: Intermittent vacuum therapy — Data on demographics and clinical conditions was gathered. The investigators collect the next features: sex, age, level of education, occupation, environment, degree of functional deficit, body mass index and Kellgren-Lawrence classification.
  Also, scores for the Knee Injury and Osteoarthritis Outcome Score, the Western Ontario and McMaster Universities Osteoarthritis Index, the Functional Independence measurement, the Fall Risk Score, and the Visual Analogue Scale were recorded at baseline and after 10 days.
  A blinded expert used a 7-15 MHz linear probe to take ultrasonographic measurements of Baker Cyst at baseline and after 10 days.
  Other Names: General warm mud bath; Hydrokinetotherapy in saline water; Massage therapy; Kinesiotherapy

SUMMARY:
The Baker cyst (BC), also known as the popliteal cyst or parameniscal cyst, is a fluid-filled sac that commonly develops in the posterior aspect of the knee, between the semimembranosus and medial head of the gastrocnemius. It is a common complication of knee osteoarthritis, and can also be associated with other conditions such as rheumatoid arthritis, gout, and meniscal tears.

BCs are typically asymptomatic, but can cause pain, stiffness, and swelling in the back of the knee. In severe cases, they can rupture, leading to inflammation and pain in the calf.

Physiotherapy is a common treatment for BCs, and has been shown to be effective in reducing size and symptoms. Intermittent vacuum therapy (IVT) is a type of physiotherapy that involves applying suction to the affected area. IVT is thought to work by increasing blood flow and lymphatic drainage, which can help to reduce inflammation and swelling.

This study aims to evaluate the effectiveness of IVT in the treatment of BCs. A total of 65 patients with knee osteoarthritis and BCs will be recruited and randomized to either a control group or an IVT group. The control group will receive standard physiotherapy treatment, while the IVT group will receive IVT in addition to standard physiotherapy treatment.

All patients will be assessed at baseline and after 10 days of treatment using a variety of clinical and functional measures, including the echo volume of the BC. The results of the study will be used to determine whether IVT is an effective treatment for BCs.

This study is designed to contribute to the existing body of knowledge on the treatment of BCs. The results of the study will be of interest to clinicians, researchers, and patients.

DETAILED DESCRIPTION:
The study was a prospective, randomized, controlled, single-blind study conducted at the Balneal and Rehabilitation Sanatorium Techirghiol (BRST) in Romania. A total of 65 patients with knee osteoarthritis (OA) and Baker's cysts (BCs) were enrolled in the study. The patients were randomly assigned to either an intermittent vacuum therapy (IVT) group or a control group.

The IVT group received IVT in addition to standard physical therapy, while the control group received standard physical therapy only. IVT was performed daily for 30 minutes using a Vacumed device. The device consists of an airtight vacuum chamber and a pump connected to a pressure control system. During vacuum treatments, participants were asked to lay themselves comfortably in a supine position. The lower body was positioned in the vacuum chamber, which was sealed around the participant's trunk with a cuff at the level of the umbilicus to allow application of negative pressure. Negative pressure cycles are created by alternating between removing air and venting the chamber to atmospheric pressure.

The standard physical therapy program consisted of a general warm mud bath (20 minutes at 38 degrees Celsius), hydrokinetotherapy in saline water from Lake Techirghiol by a certified physical therapist (20 minutes at 35 degrees Celsius), massage therapy for paravertebral muscles, shoulder and pelvis girdle, kinesio-therapy with a standard program for peripheric joints for 30 minutes.

All patients were assessed at baseline and after 10 days of treatment using a variety of clinical and functional measures, including the volume of the BC. Data on demographics and clinical conditions was gathered. The investigators collect the next features: sex, age, level of education, occupation, environment, degree of functional deficit, body mass index (BMI) and Kellgren-Lawrence classification.

Also, scores for the Knee Injury and Osteoarthritis Outcome Score (KOOS), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the Functional Independence measurement (FIM), the Fall Risk Score, and the Visual Analogue Scale (VAS) were recorded at baseline and after 10 days.

All patients were recruited at the BRST by a clinician blinded as to group allocation. Each study group was composed through random allocation of the total sample with a 1:1 allocation ratio that was reported to patients by a different researcher, who was neither the one who performed the treatment nor the one who performed the evaluation, through a pre-specified allocation list who was concealed in a password-protected computer file.

Of the total of 102 patients who were presented for hospitalization in the BRST between November and December 2022, only 65 completed the participation conditions, being grouped into two groups of 33 and 32, respectively. Due to the relatively small number of patients, the statistical approach was a non-parametric one: Independent Samples Mann Whitney U test, Independent Sample Median Test, Reb test Samples Wilcoxon Signed Rank test and Chi-Square test.

ELIGIBILITY:
Inclusion Criteria:

* free consent based on explaining and understanding all related procedural steps;
* age over 18 years;
* diagnosis of knee osteoarthritis with Baker Cyst.

Exclusion Criteria:

* neurological conditions
* rheumatological conditions
* trauma
* a history of knee or lower extremity joint surgery,
* a history of hip or ankle pain
* a history of steroid injection in the previous three months,
* conditions that would be contraindicated by Intermittent Vacuum Therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Cyst Baker Dimensions | Two measurements, on the first day of treatment and after 10 consecutive days of treatment
  Ultrasonographic measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Balneal and Rehabilitation Sanatorium Techirghiol, Techirghiol, Constanța County, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Abate M, Di Carlo L, Di Iorio A, Salini V. Baker's Cyst with Knee Osteoarthritis: Clinical and Therapeutic Implications. Med Princ Pract. 2021;30(6):585-591. doi: 10.1159/000518792. Epub 2021 Aug 2. PMID 34348320
- [Background] Henricsdotter C, Ellegaard K, Klokker L, Bartholdy C, Bandak E, Bartels EM, Bliddal H, Henriksen M. Changes in ultrasound assessed markers of inflammation following intra-articular steroid injection combined with exercise in knee osteoarthritis: exploratory outcome from a randomized trial. Osteoarthritis Cartilage. 2016 May;24(5):814-21. doi: 10.1016/j.joca.2015.12.010. Epub 2015 Dec 31. PMID 26746147
- [Background] Di Sante L, Paoloni M, Ioppolo F, Dimaggio M, Di Renzo S, Santilli V. Ultrasound-guided aspiration and corticosteroid injection of Baker's cysts in knee osteoarthritis: a prospective observational study. Am J Phys Med Rehabil. 2010 Dec;89(12):970-5. doi: 10.1097/PHM.0b013e3181fc7da2. PMID 21403593
- [Background] Zhou XN, Li B, Wang JS, Bai LH. Surgical treatment of popliteal cyst: a systematic review and meta-analysis. J Orthop Surg Res. 2016 Feb 15;11:22. doi: 10.1186/s13018-016-0356-3. PMID 26879283
- [Background] Wiecha S, Jarocka M, Wisniowski P, Cieslinski M, Price S, Makaruk B, Kotowska J, Drabarek D, Cieslinski I, Sacewicz T. The efficacy of intermittent pneumatic compression and negative pressure therapy on muscle function, soreness and serum indices of muscle damage: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2021 Nov 13;13(1):144. doi: 10.1186/s13102-021-00373-2. PMID 34774089
- [Background] Parganlija D, Nieberg V, Sauer M, Rittweger J, Bloch W, Zange J. Lower body negative pressure enhances oxygen availability in the knee extensor muscles during intense resistive exercise in supine position. Eur J Appl Physiol. 2019 Jun;119(6):1289-1303. doi: 10.1007/s00421-019-04113-w. Epub 2019 Mar 26. PMID 30915538
- [Background] Dong HH, Gao BH, Zhu H, Yang ST. [The effects of lower limb intermittent negative pressure therapy on the skin microcirculation perfusion of quadriceps in male rowers]. Zhongguo Ying Yong Sheng Li Xue Za Zhi. 2019 Feb;35(2):126-129. doi: 10.12047/j.cjap.5727.2019.028. Chinese. PMID 31250602
- [Background] Yogendrakumar V, Lun R, Hutton B, Fergusson DA, Dowlatshahi D. Comparing pharmacological venous thromboembolism prophylaxis to intermittent pneumatic compression in acute intracerebral haemorrhage: protocol for a systematic review and network meta-analysis. BMJ Open. 2018 Nov 5;8(11):e024405. doi: 10.1136/bmjopen-2018-024405. PMID 30397010
- [Background] Sarman H, Muezzinoglu US, Memisoglu K, Baran T. Vacuum-assisted closure for skin necrosis after revision total knee arthroplasty. Int Wound J. 2016 Oct;13(5):843-7. doi: 10.1111/iwj.12390. Epub 2014 Dec 30. PMID 25597628
- [Background] Hageman D, Fokkenrood HJP, van Deursen BAC, Gommans LNM, Cancrinus E, Scheltinga MRM, Teijink JAW. Randomized controlled trial of vacuum therapy for intermittent claudication. J Vasc Surg. 2020 May;71(5):1692-1701.e1. doi: 10.1016/j.jvs.2019.08.239. Epub 2019 Nov 2. PMID 31690523
- [Background] Derouet H, Caspari D, Rohde V, Rommel G, Ziegler M. Treatment of erectile dysfunction with external vacuum devices. Andrologia. 1999;31 Suppl 1:89-94. doi: 10.1111/j.1439-0272.1999.tb01456.x. PMID 10643525
- [Background] Xiang J, Wu D, Li J. Clinical Efficacy of Mudpack Therapy in Treating Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Studies. Am J Phys Med Rehabil. 2016 Feb;95(2):121-31. doi: 10.1097/PHM.0000000000000354. PMID 26203645
- [Background] Sukenik S. Balneotherapy for rheumatic diseases at the Dead Sea area. Isr J Med Sci. 1996 Jul;32 Suppl:S16-9. PMID 8756970
- [Background] Vojtassak J Jr, Vojtassak J Sr. Ultrasound monitoring of the treatment of clinically significant knee osteoarthritis. Bratisl Lek Listy. 2014;115(2):86-90. PMID 24601702
- [Background] Han DY, Ryu KN, Park JS, Jin W, Park SY, Yun SJ. The prevalence of Baker cyst in relation to the arrangement pattern between the medial head of gastrocnemius tendon and the semimembranosus tendon. Eur Radiol. 2020 Mar;30(3):1544-1553. doi: 10.1007/s00330-019-06472-6. Epub 2019 Dec 6. PMID 31811432
- [Background] Kanthawang T, Bodden J, Joseph GB, Lane NE, Nevitt M, McCulloch CE, Link TM. Obese and overweight individuals have greater knee synovial inflammation and associated structural and cartilage compositional degeneration: data from the osteoarthritis initiative. Skeletal Radiol. 2021 Jan;50(1):217-229. doi: 10.1007/s00256-020-03550-5. Epub 2020 Jul 23. PMID 32699956
- [Background] Laberge MA, Baum T, Virayavanich W, Nardo L, Nevitt MC, Lynch J, McCulloch CE, Link TM. Obesity increases the prevalence and severity of focal knee abnormalities diagnosed using 3T MRI in middle-aged subjects--data from the Osteoarthritis Initiative. Skeletal Radiol. 2012 Jun;41(6):633-41. doi: 10.1007/s00256-011-1259-3. Epub 2011 Sep 2. PMID 21887596
- [Background] Malas FU, Kara M, Kaymak B, Akinci A, Ozcakar L. Ultrasonographic evaluation in symptomatic knee osteoarthritis: clinical and radiological correlation. Int J Rheum Dis. 2014 Jun;17(5):536-40. doi: 10.1111/1756-185X.12190. Epub 2013 Oct 29. PMID 24618242
- [Background] Saylik M, Gokkus K, Sahin MS. Factors affecting Baker cyst volume, with emphasis on cartilage lesion degree and effusion in the young and middle-aged population. BMC Musculoskelet Disord. 2021 Oct 5;22(1):851. doi: 10.1186/s12891-021-04721-8. PMID 34610817
- [Background] Roos EM, Roos HP, Lohmander LS. WOMAC Osteoarthritis Index--additional dimensions for use in subjects with post-traumatic osteoarthritis of the knee. Western Ontario and MacMaster Universities. Osteoarthritis Cartilage. 1999 Mar;7(2):216-21. doi: 10.1053/joca.1998.0153. PMID 10222220
- [Background] Kandemirli GC, Basaran M, Kandemirli S, Inceoglu LA. Assessment of knee osteoarthritis by ultrasonography and its association with knee pain. J Back Musculoskelet Rehabil. 2020;33(4):711-717. doi: 10.3233/BMR-191504. PMID 31771037
- [Background] Sukenik S, Flusser D, Codish S, Abu-Shakra M. Balneotherapy at the Dead Sea area for knee osteoarthritis. Isr Med Assoc J. 1999 Oct;1(2):83-5. PMID 10731301
- [Background] Nejati P, Farzinmehr A, Moradi-Lakeh M. The effect of exercise therapy on knee osteoarthritis: a randomized clinical trial. Med J Islam Repub Iran. 2015 Feb 25;29:186. eCollection 2015. PMID 26034739
- [Background] Handy JR. Popliteal cysts in adults: a review. Semin Arthritis Rheum. 2001 Oct;31(2):108-18. doi: 10.1053/sarh.2001.27659. PMID 11590580
- [Background] Kan HS, Chan PK, Chiu KY, Yan CH, Yeung SS, Ng YL, Shiu KW, Ho T. Non-surgical treatment of knee osteoarthritis. Hong Kong Med J. 2019 Apr;25(2):127-133. doi: 10.12809/hkmj187600. Epub 2019 Mar 28. PMID 30919810
- [Background] Balik MS, Turan A, Celik FB. Is There A Relationship Between Three-Dimensionally Measured Baker's Cyst Volume and Knee Pathologies? Eurasian J Med. 2019 Feb;51(1):64-69. doi: 10.5152/eurasianjmed.2019.18385. PMID 30911260
- [Background] Eker Buyuksireci D, Buyuksireci M, Komut E. Evaluation of the effects of dexamethasone iontophoresis, galvanic current, and conservative treatment on pain and disability in patients with knee osteoarthritis and Baker's cyst. Turk J Phys Med Rehabil. 2022 Nov 22;68(4):509-516. doi: 10.5606/tftrd.2022.9213. eCollection 2022 Dec. PMID 36589359
- [Background] Manlapaz DG, Sole G, Jayakaran P, Chapple CM. Risk Factors for Falls in Adults with Knee Osteoarthritis: A Systematic Review. PM R. 2019 Jul;11(7):745-757. doi: 10.1002/pmrj.12066. Epub 2019 Mar 28. PMID 30609282
- [Background] Mat S, Tan MP, Kamaruzzaman SB, Ng CT. Physical therapies for improving balance and reducing falls risk in osteoarthritis of the knee: a systematic review. Age Ageing. 2015 Jan;44(1):16-24. doi: 10.1093/ageing/afu112. Epub 2014 Aug 22. PMID 25149678
- [Background] Park GY, Kwon DR, Kwon DG. Clinical, Radiographic, and Ultrasound Findings Between Simple and Complicated Baker's Cysts. Am J Phys Med Rehabil. 2020 Jan;99(1):7-12. doi: 10.1097/PHM.0000000000001263. PMID 31335340
- [Background] Osteras N, Kjeken I, Smedslund G, Moe RH, Slatkowsky-Christensen B, Uhlig T, Hagen KB. Exercise for hand osteoarthritis. Cochrane Database Syst Rev. 2017 Jan 31;1(1):CD010388. doi: 10.1002/14651858.CD010388.pub2. PMID 28141914
- [Background] Hautmann MG, Jung EM, Beyer LP, Suss C, Steger F, Weber M, Pohl F, Kolbl O, Putz FJ. Is low dose radiotherapy an effective treatment for Baker's cyst? Strahlenther Onkol. 2019 Jan;195(1):69-76. doi: 10.1007/s00066-018-1389-9. Epub 2018 Oct 30. PMID 30377698
- [Background] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Oo WM, Linklater JM, Bennell KL, Pryke D, Yu S, Fu K, Wang X, Duong V, Hunter DJ. Are OMERACT Knee Osteoarthritis Ultrasound Scores Associated With Pain Severity, Other Symptoms, and Radiographic and Magnetic Resonance Imaging Findings? J Rheumatol. 2021 Feb;48(2):270-278. doi: 10.3899/jrheum.191291. Epub 2020 May 15. PMID 32414954
- [Background] Bevers K, Bijlsma JW, Vriezekolk JE, van den Ende CH, den Broeder AA. The course of ultrasonographic abnormalities in knee osteoarthritis: 1 year follow up. Osteoarthritis Cartilage. 2014 Oct;22(10):1651-6. doi: 10.1016/j.joca.2014.06.012. PMID 25278074